CLINICAL TRIAL: NCT03894358
Title: Iron Absorption From a Wheat-based Instant Cereal Containing Ferrous Fumarate and Ascorbic Acid With and Without Prebiotics: Gut Microbiome and Stable Isotope Studies in Kenyan Infants
Brief Title: Iron Absorption From a Wheat-based Instant Cereal:Gut and Stable Isotope Studies in Kenyan Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: Danone Nutricia Research (Industry)
Responsible Party: Principal Investigator, Prof. Michael B. Zimmermann, Principal investigator, Swiss Federal Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INSPIRE
Record Dates: First submitted 2019-03-07; First posted 2019-03-28 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Iron Absorption; Gut Microbiota

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FeFum and 7.5 g prebiotic mixture (Active Comparator): Intervention will be 3.6 mg Fe as Ferrous Fumarate and 7.5 g of prebiotic (high dose/low dose) mixture
  Interventions: Dietary Supplement: FeFum and 7.5 g prebiotic mixture
- FeFum and 3 g prebiotic mixture (Active Comparator): Intervention will be 3.6 mg Fe as Ferrous Fumarate and 3 g of prebiotic (high dose/low dose) mixture
  Interventions: Dietary Supplement: FeFum and 3 g prebiotic mixture
- FeFum and no prebiotic mixture (Active Comparator): Intervention will be 3.6 mg Fe as Ferrous Fumarate
  Interventions: Dietary Supplement: Fefum and no prebiotic mixture

INTERVENTIONS:
Dietary Supplement: FeFum and 7.5 g prebiotic mixture — The 3 weeks intervention will consist of 24 g of wheat-based instant cereal and 90 ml of water per portion and will contain 3.6 mg FeFum and AA (molar ratio Fe:AA between 2.5 and 3) plus 7.5 g prebiotics mixture
  The absorption study test meals will consist of 24 g wheat-based instant cereal and 90 ml of water per portion and additionally:
  Test meal 1 will be composed of: 3.6 mg of Fe as 57FeFum and 0 g prebiotic mixture added extrinsically.
  Test meal 2 will be composed of: 3.6 mg of Fe as 1.5 mg iron as 58FeFum, 2.09 mg iron as 56FeFum and 7.5 g prebiotic mixture added extrinsically.
  Arms: FeFum and 7.5 g prebiotic mixture
Dietary Supplement: FeFum and 3 g prebiotic mixture — Standard wheat-based instant cereal containing 3.6 mg FeFum and AA (molar ratio Fe:AA between 2.5 and 3) plus 3 g prebiotics mixture per portion
  Arms: FeFum and 3 g prebiotic mixture
Dietary Supplement: Fefum and no prebiotic mixture — Standard wheat-based instant cereal containing 3.6 mg FeFum and AA (molar ratio Fe:AA between 2.5 and 3) per portion.
  Arms: FeFum and no prebiotic mixture

SUMMARY:
The aim of this study is to measure the effect of a prebiotic (high dose/low dose) mixture at different doses within a wheat-based instant cereal, on fractional iron absorption (FIA), gut microbiota and inflammation after three weeks. FIA will be compared with and without three weeks of pre-feeding with two different doses of the prebiotic mixture.

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) is prevalent in infants and preschool children in sub-Saharan Africa. Several studies have been conducted to mitigate IDA. Some of these studies had adverse effects on the gut microbiome and diarrhea due to the high iron dose administered in areas of high burden of malaria and other common childhood infections. As a potentially safer solution, we investigated the effect of lowering the iron dose in the iron supplements and including 7.5 g galacto-oligosaccharides (GOS). Findings from these studies demonstrated that in infants, consumption of iron and GOS improved iron status, improved the gut microbiota and reduced risk of illness. We recently demonstrated that habitual consumption of GOS for three weeks resulted in improved iron absorption that correlated with a decrease in colonic pH. It is not known whether other prebiotics or a combination will also result in increased iron absorption and what the effect of using half the dose of prebiotics would be. The composition of Human Milk Oligosaccharides (HMOs) in breast milk might be an important determinant of the gut microbiome composition and health of the breastfed infant by determining the composition of Bifidobacteria species that are the main commensal 'barrier' bacteria in the infant's gut microbiome. However, little is known about the specific HMOs composition of breast milk in African populations and the potential impact on the gut microbiota composition of the breastfed infants. We therefore aim to measure the effect of a prebiotic (high dose/low dose) mixture at different doses within a wheat-based instant cereal, on fractional iron absorption (FIA) from a wheat-based instant cereal containing no prebiotic. We will compare the FIA with and without three weeks of pre-feeding with two different doses of prebiotic mixture. In addition, we will investigate the effect of two different doses of this prebiotic (high dose/low dose) mixture on gut microbiota and inflammation after three weeks.

In south coast Kenya, we will enroll 195 infants and randomize them into three intervention groups. Daily for 3 weeks, infants will consume a newly formulated wheat-based instant cereal (3.6 mg iron with Ascorbic acid (AA)) at home. Group 1 will receive the cereal with 7.5 g prebiotic mixture; group 2 will receive the cereal with 3 g prebiotic mixture and group 3 will receive the cereal with no prebiotics. In a subset of 70 infants, we will administer four labelled test meals. Two test meals will be fed 2 weeks before beginning the intervention study to investigate the acute effect of prebiotics on FIA and the other two will be fed at the end of the 3 weeks intervention study to investigate the effect of chronic consumption of prebiotics on FIA. Breast milk samples from the mothers will be collected and analyzed for the composition of human milk oligosaccharides (HMOs). We hypothesize that: 1) Infants receiving the new wheat-based instant cereal containing prebiotic (high dose/low dose) mixture will have a higher iron absorption, and 2) higher fecal Bifidobacteria abundance than infants receiving the cereal without prebiotics; 3) in infants receiving the wheat-based instant cereal, the addition of 7.5 g of prebiotic (high dose/low dose) mixture will result in higher FIA, and 4) in greater ratio of Bifidobacteria to Enterobacteriaceae, lowest fecal calprotectin, intestinal fatty acid-binding protein (I-FABP) and lowest abundances of enteropathogens than the addition of 3 g of prebiotics; 5) the addition of 7.5 g of prebiotic (high dose/low dose) mixture will result in greater FIA when administered acutely or chronically and these two effects will be additive; 6) the wheat-based instant cereal will improve iron status, including hemoglobin (Hb), plasma ferritin (PF) and soluble transferrin receptor (sTfR), and inflammation status, including C-reactive protein (CRP), alpha-1-acid glycoprotein (AGP), fecal calprotectin and I-FABP; 7) the wheat-based instant cereal will decrease fecal pH, thereby providing a less favorable growth environment for enteric pathogens; 8) Maternal secretor status will affect the infant gut microbiota, with infants of secretor mothers having higher abundances of Bifidobacterium and Bacteroides but lower abundances of enteropathogens; and 9) Effects of co-provision of prebiotic mixture on the infant gut microbiota and on iron absorption, will be stronger among infants of non-secretor mothers.

This study will generate crucial data for optimizing iron and prebiotic-composition of wheat-based instant cereal designed for complementary feeding during infancy. This cereal could potentially be part of continued research on interventions to reduce the burden of IDA using safer formulations not adversely affecting the infant's gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 11 months at baseline
* Anticipated residence in study area for the study duration
* In good health as assessed by professional staff at Msambweni County Referral hospital
* Caregiver is willing to participate and able to comply with study procedures
* Informed consent form has been read and signed by the caregiver (or has been read out to the caregiver)

Exclusion Criteria:

* Hemoglobin concentration less than 70 g/L
* Severe underweight (Z-score weight-for-age <-3)
* Severe wasting (Z-score weight-for-height <-3
* Chronic or acute illness or other conditions that in the opinion of the Principal Investigator (PI) or study pediatrician would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol
* Participant taking part in other studies requiring the drawing of blood
* Regular intake (>2 days) of iron-containing mineral and vitamin supplements or fortified foods within the last 2 months
* Antibiotic treatment in the past 4 weeks prior to study enrollment

Ages: 6 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-01-04 (Actual); Study Completion 2020-01-04 (Actual)

PRIMARY OUTCOMES:
Fractional iron absorption (%) | Day 18
  Fractional iron absorption (erythrocyte incorporation of stable iron isotopes after 14 days of meal) from the wheat-based instant cereal containing FeFum and AA, with and without a prebiotic mixture after single dosing
Fractional iron absorption (%) | Day 57
  Fractional iron absorption (erythrocyte incorporation of stable iron isotopes after 14 days of meal) from the wheat-based instant cereal containing FeFum and AA, with and without a prebiotic mixture after long-term dosing

SECONDARY OUTCOMES:
Change in fecal Bifidobacteria abundance | Day 18 and day 39
  Dose-dependent prebiotic mediated-effect (7.5 g vs. 3 g vs. 0 g prebiotic) on fecal Bifidobacteria abundance before and after 3-week intervention
Plasma ferritin | Baseline, Day 18, Day 39, Day 57
  Iron status measured at each blood draw
Soluble transferrin receptor | Baseline, Day 18, Day 39, Day 57
  Iron status measured at each blood draw
C-reactive protein | Baseline, Day 18, Day 39, Day 57
  Inflammation status measured at each blood draw
Alpha-1-acid glycoprotein | Baseline, Day 18, Day 39, Day 57
  Inflammation status measured at each blood draw
Change in fecal calprotectin | Day 18 and Day 39
  Dose-dependent prebiotic mediated-effect (7.5 g vs. 3 g vs. 0 g prebiotic) on fecal calprotectin (inflammation marker) before and after 3-week intervention
Change in intestinal integrity | Day 18 and day 39
  An indicator of gut inflammation; assessed by measuring Intestinal fatty acid binding protein (I-FABP) in fecal samples; Dose-dependent prebiotic mediated-effect (7.5 g vs. 3 g vs. 0 g prebiotic) before and after 3-week intervention
Change in gut microbiome composition | Day 18 and day 39
  Change in composition of the gut microbiome including pathogens; Dose-dependent prebiotic mediated-effect (7.5 g vs. 3 g vs. 0 g prebiotic) before and after 3-week intervention, assessed using qPCR, metagenomics and 16s sequencing
Change in fecal pH | Day 18 and Day 39
  Dose-dependent prebiotic mediated-effect (7.5 g vs. 3 g vs. 0 g prebiotic) before and after 3-week intervention
Short chain fatty acids concentrations | Day 18 and day 39
  Dose-dependent prebiotic mediated-effect (7.5 g vs. 3 g vs. 0 g prebiotic) before and after 3-week intervention
Change in viral load in nasopharynx | Day 18 and day 39
  Potential upper respiratory tract pathogens will be assessed in the nasopharyngeal swabs collected; Dose-dependent prebiotic mediated-effect (7.5 g vs. 3 g vs. 0 g prebiotic) before and after 3-week intervention
Maternal secretor status and HMO concentrations | Day 39
  HMO concentrations in the breast milk of the mothers of the participating infants will be measured on day 39 and the maternal secretor status will be determined.
  Effect of maternal secretor status on the infant gut microbiota and response to iron fortificants with or without co-provision of prebiotics will be investigated

CONTACTS AND LOCATIONS:
Locations (1):
- Msambweni County Referral Hospital, Msambweni, Kwale County, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mikulic N, Uyoga MA, Stoffel NU, Derrien M, Nyilima S, Kostopoulos I, Roeselers G, Chenoll E, Mwasi E, Pironaci G, Karanja S, Bourdet-Sicard R, Zimmermann MB. Prebiotics increase iron absorption and reduce the adverse effects of iron on the gut microbiome and inflammation: a randomized controlled trial using iron stable isotopes in Kenyan infants. Am J Clin Nutr. 2024 Feb;119(2):456-469. doi: 10.1016/j.ajcnut.2023.11.018. Epub 2023 Nov 30. PMID 38042412
- [Derived] Derrien M, Mikulic N, Uyoga MA, Chenoll E, Climent E, Howard-Varona A, Nyilima S, Stoffel NU, Karanja S, Kottler R, Stahl B, Zimmermann MB, Bourdet-Sicard R. Gut microbiome function and composition in infants from rural Kenya and association with human milk oligosaccharides. Gut Microbes. 2023 Jan-Dec;15(1):2178793. doi: 10.1080/19490976.2023.2178793. PMID 36794816